CLINICAL TRIAL: NCT00965380
Title: A Radiographic and Clinical Study Evaluating a Novel Allogeneic, Cancellous, Bone Matrix Containing Viable Stem Cells (Trinity Evolution™ Viable Cryopreserved Cellular Bone Matrix) in Posterior Lumbar or Transforaminal Lumbar Interbody Fusion (PLIF or TLIF)
Brief Title: Trinity Evolution in Posterior or Transforaminal Lumbar Interbody Fusion (PLIF/TLIF)
Acronym: TLF
Status: Completed | Type: Observational
Sponsor: Orthofix Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-01006B
Record Dates: First submitted 2009-08-21; First posted 2009-08-25 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Degenerative Disc Disease
Keywords: Trinity Evolution; Symptomatic lumbar degenerative disc disease; Posterior lumbar interbody fusion; Transforaminal lumbar interbody fusion
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to utilize Trinity Evolution in conjunction with an interbody spacer and supplemental posterior fixation of the surgeon's choice and to follow the patients to measure the clinical outcomes and rate of fusion. The hypothesis of the study is that Trinity Evolution combined with an interbody spacer and supplemental posterior fixation will result in fusion rates and clinical outcomes similar to those with other routinely used autograft and allograft materials including: fusion, improvement in pain and function, maintenance of lower extremity neurological function, and absence of serious adverse events related to the use of the Trinity Evolution product.

DETAILED DESCRIPTION:
Degenerative disorders of the lumbar spine can lead to a multitude of clinical problems including back pain and/or leg pain secondary to nerve compression and/or deformity. When conservative (non-surgical) treatment fails after at least a 6 month period and/or non-operative treatment is not indicated, patients and physicians may turn to a surgical solution. Surgical options consist basically of decompressing nerves, correcting and/or stabilizing deformities if required and fusing the segment, depending on the clinical situation. The "gold standard" for aiding healing in spinal fusion surgeries is the harvesting of autograft from the patient's iliac crest and placing it in and around the segments of the spine that are intended to be fused. Autograft is considered the "gold standard" because it contains the essential elements required for successful bone grafting: osteogenesis, osteoconduction, and osteoinduction.

However, the morbidity of harvesting autograft has been well documented and includes chronic donor-site pain, infection, neurologic injury, blood loss, deformity, bowel injury, hernia, and prolonged surgical and hospitalization time. There are now a number of products on the market to minimize or replace the use of autograft. However, few of these products contain all three essential bone-forming elements (osteogenesis, osteoconduction, and osteoinduction) in a single, stand alone product.

Trinity Evolution is a novel, allogeneic cancellous bone matrix containing viable osteoprogenitor cells, mesenchymal stem cells and a demineralized cortical bone (DCB) component to provide the required osteoconduction, osteogenesis, and osteoinduction necessary for successful bone grafting. Preclinical studies with Trinity Evolution have demonstrated in-vitro and in-vivo safety and effectiveness. Trinity Evolution is considered an allograft and as such is a "minimally manipulated" tissue and is labeled for bone repair for spinal, orthopedic and podiatric indications where autograft is used. The dosage will be dependent upon the specific requirements of the case.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic lumbar degenerative disc disease at 1 or 2 adjacent levels between L3 and S1
* Patients with back and/or leg pain scheduled for stabilization with or without decompression via a TLIF or PLIF approach utilizing an interbody spacer and supplemental posterior fixation.
* Greater than 18 years of age
* Unresponsive to conservative care over a period of at least 6 months or has progressive neurological signs and/or symptoms of neurological compromise that mandate urgent surgical intervention
* Willing and able to comply with the requirements of the protocol including follow-up requirements
* Willing and able to sign a study specific informed consent.

Exclusion Criteria:

* Patients requiring surgical treatment other than at 1 or 2 adjacent levels between L3 and S1
* Active local or systemic infection
* Currently pregnant or considering becoming pregnant during the follow-up period
* Active malignancy or having been on chemotherapy of any kind for a malignancy in the past 1 year
* Use of any other bone graft or bone graft substitute in addition to or in place of Trinity Evolution matrix in and around the interbody spacer.
* Use of adjunctive post-operative stimulation
* Prior interbody surgery at the same level
* Has a known history of hypersensitivity or anaphylactic reaction to dimethyl sulfoxide (DMSO).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic lumbar degenerative disc disease scheduled to undergo PLIF or TLIF.
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2009-09; Primary Completion 2014-11 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Fusion Rates for Trinity Evolution | Operative to 24 months follow-up

SECONDARY OUTCOMES:
NDI relative improvement; VAS improvement; Maintenance or improvement of neurological function | Pre-op to 24 months follow-up
Complication Rates for Trinity Evolution | Operative to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: James T Ryaby, PhD, Study Director — Orthofix Inc.
Locations (15):
- United States (15):
  - Boulder Neurosurgical Associates, Boulder, Colorado
  - Total Spine Care, Canton, Connecticut
  - Middlesex Orthopedic Surgeons, Middletown, Connecticut
  - Center for Advanced Neuro and Spine, New Britain, Connecticut
  - Optim Healthcare (Formerly Southeastern Orthopedic Center), Savannah, Georgia
  - Parkview Orthopaedic Group, Palos Heights, Illinois
  - Willis Knighton Health System, Shreveport, Louisiana
  - University of Michigan A. Alfred Taubman Health Care Center, Ann Arbor, Michigan
  - Cooper University Neurological Institute, Camden, New Jersey
  - Spine Surgery of Buffalo Niagara, Niagara Falls, New York
  - Carolina NeuroSurgery & Spine, Charlotte, North Carolina
  - Triangle Orthopaedic Associates, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - Triangle Neurosurgery, Raleigh, North Carolina
  - Tuckahoe Orthopedic Surgeons, Richmond, Virginia